CLINICAL TRIAL: NCT03894488
Title: Clinical Evaluation of the Application of the FilmArray GI Panel in Post-HSCT
Brief Title: Clinical Evaluation of the Application of the FilmArray GI Panel in Post-HSCT Diarrhea Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Principal Investigator, Cao Qing, Director of Infectious Diseases, Shanghai Children's Medical Center
Other Study IDs: GI-GVHD
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: GVHD - Graft-Versus-Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FilmArray Gastrointestinal (GI) Panel — The FilmArray GI Panel tests for 22 of the most commonly associated pathogens related to gastroenteritis-all from one patient sample, one easy to use reagent, and results are available in about one hour.

SUMMARY:
This is a prospective single arm study with the study period from June 1st, 2019 to May 31st, 2020. An historical control group will be used in the study, which includes all patients received HSCT but not GI panel detection between June 1st, 2018 to May 31st, 2019. All patients receiving HSCT within the year at SCMC will be enrolled in the study. The stool samples will be collected from each patient at 2-3 time points, including the day before pre-conditioning (T1), 28+-3 days after HSCT (T2), and the day severe diarrhea present (T3). All the stool samples will be detected by the FilmArray GI panel, and the results as well as other clinical information including the laboratory examinations will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years old;
* Receiving HSCT;
* Legal guardians fully understand and sign informed consent.

Exclusion Criteria:

* Receiving secondary transplantation;
* Cannot give informed consent or not willing to enroll the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients receiving HSCT within the year at SCMC
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive rate of FilmArray GI test before and post-HSCT | 31 days after HSCT
Compare the FilmArray GI test results generated from the same patients in different time points | 31 days after HSCT

IPD SHARING:
Plan to Share IPD: Undecided